CLINICAL TRIAL: NCT00727168
Title: Epidemiologic Study for the Prevalence of Glaucoma in Namil Area, Geumsan City, South Korea
Brief Title: Screening for Glaucoma in Namil Area, South Korea
Status: Completed | Type: Observational
Sponsor: Korean Glaucoma Society (Network)
Responsible Party: Gong-je Seong, president, Korean Glaucoma Society
Other Study IDs: CNUH81510-9701
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Last update posted 2008-08-04 (Estimated); Status verified 2008-08

CONDITIONS: Glaucoma; Intraocular Pressure; Optic Nerve Head; Visual Field
Keywords: prevalence study; glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to study the prevalence of glaucoma in Korea, the investigators selected Namil area in Geumsan city, located in central Korea. The residents aged over 40 in this area are to be recruited to full ophthalmologic examination to detect and classify the glaucoma.

DETAILED DESCRIPTION:
Screening includes following examinations; Questionaire and Consent form, Visual acuity test, Auto-refraction, IOL Master measurement, Pachymetry, FDT Perimetry, Fundus Photography, Slit lamp examination, Goldmann applanation Tonometry, Gonioscopy, and Binocular optic disc evaluation. For the cases showing any abnormality in FDT perimetry, optic disc morphology, or intraocular pressure, Humphrey automated visual field test is to be performed as an extended examination. Finally, optic nerve head evaluation by OCT or GDx analyzer is to be used as a confirmation test, as well as additional Humphrey visual field test.

ELIGIBILITY:
Inclusion Criteria:

* All residents aged over 40 in Namil area

Exclusion Criteria:

* Individuals registered but not actually living in this area

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All residents aged over 40 in Namil area in Geumsan city
Sampling Method: Probability Sample
Enrollment: 1532 (Actual)
Dates: Start 2007-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Prevalence of glaucoma in Namil area | cross-sectional

SECONDARY OUTCOMES:
Clinical factors associated with the glaucoma | cross-sectional

CONTACTS AND LOCATIONS:
Overall Officials: Gong-je Seong, MD, PhD, Principal Investigator — Korean Glaucoma Society
Locations (1):
- Yongdong Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim YY, Lee JH, Ahn MD, Kim CY; Namil Study Group, Korean Glaucoma Society. Angle closure in the Namil study in central South Korea. Arch Ophthalmol. 2012 Sep;130(9):1177-83. doi: 10.1001/archophthalmol.2012.1470. PMID 22965594